CLINICAL TRIAL: NCT03726450
Title: Can Myo-inositol in Combination With N-Acetyl-Cysteine Plus an Antioxidant Mix be Useful for the Management of Men Affected by Idiopathic Infertility and Semen Hyperviscosity?
Brief Title: Myo-inositol and an Antioxidant Mix for the Treatment of Vietnamese Infertile Men
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Andrology and Fertility Hospital of Hanoi (Other)
Responsible Party: Principal Investigator, Hung Nguyen Ba, Andrologist, Andrology and Fertility Hospital of Hanoi
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAVIM
Record Dates: First submitted 2018-09-07; First posted 2018-10-31 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-03

CONDITIONS: Male Infertility
Keywords: myo-inositol; N-acetyl-cysteine; semen hyperviscosity; idiopathic male infertility
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Andrositol Plus (Experimental): all the patients will be treated for three months with a dietary supplement containing Myo-inositol, NAC, Folic acid, selenium, vitamin E, L-Arginine and L-Carnitine
  Interventions: Dietary Supplement: Andrositol Plus

INTERVENTIONS:
Dietary Supplement: Andrositol Plus — Myo-inositol
Dietary Supplement: Andrositol Plus — N-Acetyl-Cysteine
Dietary Supplement: Andrositol Plus — Folic Acid
Dietary Supplement: Andrositol Plus — Selenium
Dietary Supplement: Andrositol Plus — L-arginine
Dietary Supplement: Andrositol Plus — L-carnitine
Dietary Supplement: Andrositol Plus — Vitamin E

SUMMARY:
The aim of this study is to evaluate if Myo-inositol, N-Acetyl-Cysteine plus a cocktail of antioxidants could be able to increase spermatozoa parameters and reduce semen hyper-viscosity

DETAILED DESCRIPTION:
According to the World Health Organization (WHO), the incidence of infertile couples is relatively high, with a range from 15% to 20% in the developed countries. In accordance with WHO, spermatogenesis disorders occur in almost 50% of all the cases of male infertility. In the recent decades, an unexplained reduction has been found, not only in sperm quality and quantity but also in the volume of the ejaculate. This evidence allows speculations on the number of male infertility factors, which will keep increasing in the future. An important impact on male infertility caused by environmental factors, such as bad habits (alcohol and smoking), body overload and in particular the reluctance of men undergoing prevention is widely reported. A reduced fertility is often related to a lower sperm motility. Over the recent years, the percentage of motile sperms in the ejaculate is constantly reducing. For these reasons, WHO, in the latest edition, indicated a percentage of sperms progressive motility less than 32% as a parameter of the reduced chance of getting pregnant spontaneously. The etiopathogenesis of male infertility is extremely complex, and the factors and processes causing these disorders in the reproduction are different. A common cause of reduced sperms motility seems to be related to the toxic action of reactive oxygen species (ROS). Pathological effects of free radicals in the male reproductive tract are associated with DNA fragmentation, lipid peroxidation, and apoptosis, and these lead to reduced fertility and miscarriages. Due to this evidence, antioxidant species were introduced in the management of male infertility. Between these molecules, Selenium and L-Arginine had shown a strong impact in contrasting ROS generation and restoring the oxidative status of the seminal environment. Myo-inositol (MI) is an isomer of the inositol's family. In nature are present 9 isomers of this sugar-like and MI represents the most abundant one. It plays a key role in more than one cellular pathways as FSH, insulin and TSH second intracellular messenger. It has been also demonstrated an important effect of MI in improving semen parameters such as motility, morphology, and quality, both in vitro and in vivo. From the reported studies, the effect of this isomer seems to be related to an improvement in the membrane potential of spermatozoa's mitochondria and in the reduction of the semen amorphous material that frequently impairs male fertility. Based on this evidence, recent scientific researches have been focused on the clinical use of MI in the management of male infertility caused by semen alterations. A further growing issue impairing male fertility is semen hyperviscosity (SHV). SHV is a condition that can seriously impair the physical and chemical characteristics of the seminal fluid and it can have a serious impact on sperm function. Worth of spreading, SHV seems to be associated with reduced sperm motility, possibly due to a 'trapping effect' that prevents normal sperm progression through the female genital tract. N-acetyl-L-cysteine (NAC) is a derivative of the naturally occurring amino acid L-cysteine that has free radical scavenging activity and it is also commonly used as a mucolytic agent. In addition to NAC antioxidant activity, Cifci et al. found it effective in reducing semen viscosity and its oxidative status as well as in increasing semen volume and spermatozoa motility.

ELIGIBILITY:
Inclusion Criteria:

* BMI < 29
* One year of unsuccessful sexual intercourses without achieving pregnancy for male factor (idiopathic infertility)
* Normospermia, isolated asthenozoospermia and/or oligoasthenozoospermia
* Semen hyper-viscosity defined as severe, moderate and mild

Exclusion Criteria:

* The absence of spermatozoa production
* Positive presence of leucocyte and inflammation factor in the seminal fluid
* Positive urea test for the presence of bacteria, protozoa and/or fungi infection
* Diagnosis of cryptorchidism
* Diagnosis of Varicocele of grade 2 or higher
* Diagnosis of Diabetes and other pathology causing oxidative stress
* Concentration alterations of the following hormones: LH, FSH, Testosterone, Prolactin, 17b-estradiol
* Abuse of alcohol and controlled substance
* Smoking cigarettes (>10 cigarettes/day)
* BMI > 30

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 55 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-02-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
change in sperm motility | spermatozoa motility will be analyzed after 3 months of treatment
  spermatozoa motility will be evaluated through microscopical evalutation

SECONDARY OUTCOMES:
change in sperm morphology | spermatozoa morphology will be analyzed at the enrollment and after 3 months of treatmentanalyzed
  spermatozoa morphology will be evaluated through microscopical evalutation
change in sperm vitality | spermatozoa vitality will be analyzed after 3 months of treatment
  spermatozoa vitality will be evaluated through vitality test with methylene blue
change in sperm count | spermatozoa count will be 3 months of treatment
  spermatozoa count will be evaluated through microscopical evalutation
change in seminal fluid viscosity | semen Hyper-viscosity will be analyzed after 3 months of treatment
  Viscosity will be determined after ejaculation by gently aspirating semen into a 5 ml pipette and then producing semen drops.

CONTACTS AND LOCATIONS:
Locations (1):
- Hung Nguyen, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided